CLINICAL TRIAL: NCT07404488
Title: Prospective Randomized Controlled Study Comparing Dentoalveolar, Skeletal, Periodontal and Nasal/Airway Effects of a Two-miniscrew Bone-borne Expander, a Four-miniscrew Bone-borne Expander, and a Conventional Tooth-borne Hyrax Expander in Adolescents.
Brief Title: Comparison of Two Miniscrew Bone-borne Expanders (2 vs 4 Screws) Versus Conventional Hyrax Expander in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michele Cassetta, Professor, DDS, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS_RME
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Orthodontic Appliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Group A) - Two-miniscrew bone-borne expander (Experimental): one-borne rapid maxillary expander anchored on two palatal miniscrews inserted in paramedian palatal vault (near first-second premolar area). Miniscrews: self-tapping titanium (Benefit system; PSM Medical Solutions). Placement planned via CBCT-guided CAD/CAM surgical guide (Easy Driver). Activation protocol: Hyrax click 10 mm screw: 4 quarter-turns at placement then 3 quarter-turns/day for 12 days (0.20 mm/turn) until ~8 mm expansion.
  Interventions: Device: Miniscrew supported expander application
- Arm 2 (Group B) - Four-miniscrew bone-borne expander (Experimental): Bone-borne rapid maxillary expander anchored on four palatal miniscrews (two paramedian + two parapalatine). Same guided insertion workflow and activation protocol as Group A.
  Interventions: Device: 4 miniscrews supported rapid maxillary expansion application
- Arm 3 (Group C) - Conventional tooth-borne Hyrax expander (Active Comparator): Tooth-borne Hyrax expander banded on upper first permanent molars (conventional Hyrax). Same activation protocol as Groups A/B.
  Interventions: Device: Conventional tooth-borne Hyrax expander (comparator)

INTERVENTIONS:
Device: Miniscrew supported expander application — Two palatal miniscrews with custom bone-borne expansion framework (device transmits forces to palatal bone; no tooth bands).
  Arms: Arm 1 (Group A) - Two-miniscrew bone-borne expander
Device: 4 miniscrews supported rapid maxillary expansion application — Four palatal miniscrews with custom bone-borne expansion appliances.
  Arms: Arm 2 (Group B) - Four-miniscrew bone-borne expander
Device: Conventional tooth-borne Hyrax expander (comparator) — Hyrax-type tooth-borne expander with bands cemented on upper first molars (Hyrax click 10 mm).
  Arms: Arm 3 (Group C) - Conventional tooth-borne Hyrax expander

SUMMARY:
Rapid maxillary expansion (RME) is used to correct transverse deficiencies of the maxilla. This randomized controlled trial compares three RME devices in adolescents (age 10-15) with at least 8 mm maxillary transverse deficiency: (1) bone-borne expander supported by two palatal miniscrews, (2) bone-borne expander supported by four palatal miniscrews, and (3) conventional tooth-borne Hyrax expander. Devices were placed using static computer-guided miniscrew insertion (where applicable). All participants received the same activation protocol to reach 8 mm expansion. Cone-beam CT scans were obtained pre-treatment (T0) and at 6 months post-treatment (T1). The trial assesses skeletal, dentoalveolar, periodontal, and nasal/airway outcomes. Enrollment: 36 subjects. Study sites: Sapienza University of Rome.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel-group clinical trial performed at the Department of Oral and Maxillofacial Sciences, Sapienza University of Rome (Nov 2021 - Sep 2024). Inclusion criteria included age under 16 years, late mixed or permanent dentition, and maxillary transverse deficiency ≥ 8 mm. Exclusion: poor oral hygiene; previous orthodontic treatment; craniofacial syndromes; cleft lip/palate; genetic/congenital diseases. After consent, eligible participants (N=36) were randomized (1:1:1) to: Group A - two-miniscrew bone-borne expander (paramedian screws near 1st-2nd premolar region); Group B - four-miniscrew bone-borne expander (two paramedian + two parapalatine); Group C - Hyrax tooth-borne expander banded to upper first molars. Miniscrews (Benefit system; PSM Medical Solutions) were placed using a CAD-CAM surgical guide planned from CBCT and digital models (Easy Driver). Activation: Hyrax click 10 mm screw; four quarter-turns at insertion then three quarter-turns/day for 12 days (0.20 mm/turn; ~0.6 mm/day) until 8 mm achieved. CBCT scan acquisition: Scanora 3Dx (Soredex). Measurements performed on Simplant v17 on defined landmarks (MaxBas, MaxAlv, MaxAlvPre, Ns, ZigMax, IntermCo, IntermoAp, molar angles, periodontal bone thickness measures, nasopalatine foramen width). Primary outcome: change in maxillary basal width (MaxBas) T0 to T1 measured on CBCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 to 15 years (under 16 at enrollment).
* Late mixed or permanent dentition.
* Maxillary transverse deficiency ≥ 8 mm (unilateral or bilateral).
* Parent/guardian able to provide written informed consent; participant assent where applicable.

Exclusion Criteria:

* Poor oral hygiene.
* Prior orthodontic treatment.
* Craniofacial syndromes.
* Cleft lip and/or palate.
* Genetic or congenital diseases likely to affect craniofacial growth or bone quality.
* Inability/unwillingness to attend scheduled follow-up visits.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in maxillary basal width (MaxBas) from baseline (T0) to 6 months post-treatment (T1) | at 6 months
  Measurement method: CBCT (Simplant software) distance between alveolar/basal points (points 5-6 as per Podesser/Garib protocol).

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Rm, Italy

IPD SHARING:
Plan to Share IPD: No